CLINICAL TRIAL: NCT06252545
Title: PROmoting CLinicAl TrIal EngageMent for Pancreatic Cancer App Study (PROCLAIM Study
Brief Title: Promoting CT Engagement for Pancreatic Cancer With App
Acronym: PROCLAIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Lustgarten Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: LCCC2234
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Pancreas Cancer
Keywords: ethnicity; black; application
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: There will be 2 groups: 20 subjects with pancreas carcinoma for phone interviews and 6 for user testing the first version of the application..
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interview Group (Other): Subjects with pancreatic carcinoma who joined the interview group.
  Interventions: Behavioral: semistructured interviews
- User Testing Group (Other): Subjects with pancreatic carcinoma who joined the user testing group
  Interventions: Behavioral: feedback

INTERVENTIONS:
Behavioral: semistructured interviews — Black subjects with pancreatic cancer will provide insight on their experience discussing clinical trials and preferences for communicating clinical trial information
  Arms: Interview Group
Behavioral: feedback — Black subjects with pancreatic cancer will provide feedback on mHealth app prototype.
  Arms: User Testing Group

SUMMARY:
To develop a culturally tailored informational mobile application and test whether it will increase participation among Black pancreatic cancer subjects in clinical trial discussions with their care team.

This project aims to identify and address barriers to enrollment of Black subjects in pancreatic cancer clinical trials using a culturally informed mobile health application to promote participation.

The clinical trial education and communication needs of Black people with pancreatic cancer will be determined. A new mHealth application for clinical trial education and communication tailored to subject needs will be developed. It was hypothesized that a culturally tailored informational mobile application will increase the participation of Black subjects in clinical trial discussions with their care team among the target population.

This study focuses on Black pancreatic cancer subjects, who experience higher mortality rates and lower clinical trial participation than White subjects. Research shows that the disparity between clinical trial participation is in part due to inequitable recruitment practices. This study will use mobile application technology (mHealth app) as an educational, communication, audit, and feedback tool to promote patient-initiated clinical trial discussions among Black people with pancreatic cancer and their cancer care team.

ELIGIBILITY:
Inclusion Criteria

Participants must meet the following inclusion criteria in order to participate in communication & education interview component of the study:

1. Informed consent obtained to participate in the study
2. 18 years or older
3. English speaking
4. Able and willing to participate in a 1-hour interview
5. History of pancreatic cancer diagnosis
6. Identify as Black

Exclusion Criteria:

All participants meeting any of the following exclusion criteria will be excluded from the study:

1. Inability to read and speak English
2. Dementia altered mental status, or any psychiatric condition that would prohibit understanding or rendering of informed consent as determined by the study physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
The clinical trial education and communication needs | Up to 1 month
  The clinical trial education and communication needs of Black people with pancreatic cancer will be determined with feedback and qualitative analysis of findings from semi-structured interviews to develop an mHealth application.

CONTACTS AND LOCATIONS:
Overall Officials: Jen J Yeh, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (2):
- United States (2):
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Medical College Of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials